CLINICAL TRIAL: NCT04134468
Title: UPCC 10219: Phase II Study Of Stromal Changes Detected By DCE- and DW-MRI In Response To PEGPH20 Combined With Chemotherapy In Subjects With Locally-Advanced Pancreatic Cancer
Brief Title: MRI Effects of Pegvorhyaluronidase Alfa (PEGPH20) in Pancreatic Ductal Adenocarcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Halozyme halted development of PEGPH20 following Phase 3 failure.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC10219; IRB833642 (Other: Abramson Cancer Center)
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — PEGPH20; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegvorhyaluronidase alfa plus Abraxane and Gemcitabine (Experimental): Pegvorhyaluronidase alfa 3ug/kg IV twice weekly during Cycle 1 and then weekly on days of chemotherapy during Cycles 2-4. Abraxane 125mg/m2 IV and Gemcitabine 1000mg/m2 IV on Day 1, 8, 15 of Cycles 1-4. All cycles will be 28 days.
  Interventions: Drug: Pegvorhyaluronidase alfa; Drug: Abraxane; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pegvorhyaluronidase alfa — IV infusion
  Other Names: PEGPH20
Drug: Abraxane — IV infusion
Drug: Gemcitabine — IV infusion

SUMMARY:
This research study is being conducted to determine the effects of PEGPH20 plus chemotherapy treatment on the MRI characteristics of locally advanced pancreatic cancer patient tumors. Subjects will received Gemcitabine, Abraxane and PEGPH20.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Capable of giving informed consent.
3. Ability and willingness to comply with the protocol including all scheduled MRI studies and paired tumor biopsies
4. Aged ≥ 18 years.
5. borderline or unresectable pancreatic adenocarcinoma without distant metastatic disease.
6. ECOG PS of 0 or 1
7. Must have adequate organ and hematopoietic function
8. Female and Males must use an approved contraceptive method

Exclusion Criteria:

1. Received prior therapy for pancreatic adenocarcinoma
2. History of deep vein thrombosis (DVT) or pulmonary embolism (PE)
3. Contraindication to therapeutic anticoagulation or heparin
4. Intolerance to dexamethasone
5. Contraindication to MRI or unwillingness to undergo all scheduled MRI exams
6. Known or suspected brain metastasis
7. Significant cardiovascular disease such as current New York Heart Associate Class III/IV heart failure, myocardial infarction or stroke within 6 months prior to enrollment
8. A second primary malignancy that, in the judgment of the investigator, may affect the interpretation of results
9. Any illness or condition that in the opinion of the investigator may affect the safety of the subject or the evaluation of any study endpoint
10. Active bacterial or fungal infection requiring IV therapy at the start of protocol treatment
11. Subjects may not receive concomitant anticancer agents or radiation.
12. Female subjects who are pregnant or nursing
13. Pre-existing peripheral neuropathy > CTCAE Grade 2.
14. Known allergy to hyaluronidase
15. Current use of megestrol acetate (use within 10 days of Day 1)
16. Inability to comply with study and follow-up procedures as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-02-11 (Estimated); Study Completion 2022-11-11 (Estimated)

PRIMARY OUTCOMES:
Change in lesion size | baseline and 4 months
  Change in lesion size

SECONDARY OUTCOMES:
Proportion of patients achieving a complete R0 surgical resection | at time of surgery
  Proportion of patients achieving a complete R0 surgical resection

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Karasic, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No